CLINICAL TRIAL: NCT01458301
Title: A Phase II, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of the Efficacy and Safety of TAK-385 10, 20, and 40 mg (p.o.) in the Treatment of Endometriosis
Brief Title: Efficacy and Safety of TAK-385 in the Treatment of Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-385/CCT-101; U1111-1123-6890 (Registry Identifier: WHO); JapicCTI-111588 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-08-31; First posted 2011-10-24 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Endometriosis
Keywords: Drug Therapy
MeSH Terms: conditions — Endometriosis | interventions — relugolix; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TAK-385 10 mg QD (Experimental)
  Interventions: Drug: TAK-385
- TAK-385 20 mg QD (Experimental)
  Interventions: Drug: TAK-385
- TAK-385 40 mg QD (Experimental)
  Interventions: Drug: TAK-385
- Leuplin (Other)
  Interventions: Drug: Leuprorelin acetate

INTERVENTIONS:
Drug: Placebo — TAK-385 placebo-matching tablets, orally, once daily and Leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks.
  Arms: Placebo
Drug: TAK-385 — TAK-385 10 mg, tablets, orally, once daily and Leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks
  Arms: TAK-385 10 mg QD
Drug: TAK-385 — TAK-385 20 mg, tablets, orally, once daily and Leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks
  Arms: TAK-385 20 mg QD
Drug: TAK-385 — TAK-385 40 mg, tablets, orally, once daily and Leuprorelin acetate placebo injection, subcutaneously, once every 4 weeks for up to 12 weeks
  Arms: TAK-385 40 mg QD
Drug: Leuprorelin acetate — TAK-385 placebo-matching tablets, orally, once daily and Leuprorelin acetate injection, subcutaneously, once every 4 weeks for up to 12 weeks
  Other Names: Leuplin
  Arms: Leuplin

SUMMARY:
The purpose of this study is to determine the efficacy and safety of TAK-385, once daily (QD), for 12 weeks in women with endometriosis.

DETAILED DESCRIPTION:
This Phase II, multicenter, double-blind, randomized, parallel-group, placebo-controlled study will evaluate the efficacy and safety of 3 dose levels (10, 20, and 40 mg) of TAK-385 following oral administration for 12 weeks in women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women
2. The participants must have dysmenorrhea and pelvic pain associated with endometriosis.
3. The participant has experienced a regular menstrual cycle.
4. The participant has been diagnosed with endometriosis by method a), b), or c).

   * Laparotomy
   * Laparoscopy
   * Chocolate cyst of the ovary confirmed by MRI

Exclusion Criteria:

1. Participants diagnosed with measurable uterine fibroids with the longest diameter of 3 cm or larger
2. Participants with lower abdominal pain due to irritable bowel syndrome or severe interstitial cystitis
3. Participants with a previous or current history of thyroid dysfunction
4. Participants with current or previous history of pelvic inflammatory disease
5. Participants with positive PAP smear test result conducted
6. Participants with a history of panhysterectomy or bilateral oophorectomy
7. Participants judged by investigator to have marked abnormal uterine bleeding or anovulatory bleeding
8. Participants with a previous or current history of a malignant tumor
9. Participants who have been treated with any of the following drugs: anticoagulant drug, antiplatelet drug, tranexamic acid, selective estrogen receptor modulator (SERM), activated vitamin D, other vitamin D, calcitonin, ipriflavone, steroid hormone, vitamin K, teriparatide,or denosumab
10. Participants who have been treated with any of the following drugs: oral contraceptive and sex hormone preparation, gonadotropin-releasing hormone (GnRH) analogue, dienogest, danazol, or aromatase inhibitor
11. Participants who have been treated with bisphosphonate preparation
12. Participants with a previous or current history of hypersensitivity or allergy to Leuplin, synthetic LH-RH, LH-RH derivatives, gelatin-containing formulations or food containing gelatin, or have a previous or current history of severe hypersensitivity or severe allergy to other drugs
13. Participants with non-diagnosable abnormal genital bleeding
14. Participants with a previous or current history of osteoporosis, bone mass loss, or other metabolic bone diseases
15. Participants with clinically significant cardiovascular disease or uncontrollable hypertension
16. Participants judged by investigator to be inappropriate to participate in this study based on the 12-lead electrocardiogram (ECG) findings
17. Participants with active liver disease or jaundice, or with alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin > 1.5 times the upper limit of normal (ULN) in the clinical laboratory tests

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Score for pelvic pain as measured by the Visual Analogue Scale (VAS) | Week 12 (one menstrual cycle)
  Pelvic pain will be assessed using the VAS as pain evaluation scale.

SECONDARY OUTCOMES:
VAS Score for Pelvic Pain | Up to Week 12.
  Pelvic pain will be assessed using the VAS as pain evaluation scale
VAS Score for Dyspareunia | Up to Week 12.
  Dyspareunia will be assessed using the VAS as pain evaluation scale
Bone Mineral Density | Up to Week 12.
  Measured by Dual-energy X-ray absorptiometry (DXA)
Treatment-emergent Adverse Events. | Up to Week 16
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through the last visit (Week 16)
Vital Signs | Up to Week 12.
  Vital signs will include body temperature, sitting blood pressure and pulse (bpm).
Body Weight | Up to Week 12.
Electrocardiograms. | Up to Week 12.
Number of Participants with Markedly Abnormal Standard Safety Laboratory Values | Up to Week 24
Serum NTx | Up to Week 12.
  NTx is one of the biochemical bone metabolism markers
Serum BAP | Up to Week 12.
  BAP is one of the biochemical bone metabolism markers

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Takeda
Locations (69):
- Japan (69):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Funabashi-shi, Chiba
  - Ichihara-shi, Chiba
  - Yachiyo-shi, Chiba
  - Nihama-shi, Ehime
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Iizuka-shi, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Yanagawa-shi, Fukuoka
  - Koriyama-shi, Fukushima
  - Takayama-shi, Gifu
  - Takasaki-shi, Gunma
  - Hirosima-shi, Hiroshima
  - Ebetsu-shi, Hokkaido
  - Ishikari-shi, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kako-gun, Hyōgo
  - Kawanishi-shi, Hyōgo
  - Kobe, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Marugame-shi, Kagawa-ken
  - Kagoshima, Kagoshima-ken
  - Hiratsuka-shi, Kanagawa
  - Kamakura-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Yamato-shi, Kanagawa
  - Yokohama, Kanagawa
  - Nankoku-shi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Matsumoto-shi, Nagano
  - Nagano, Nagano
  - Suzaka-shi, Nagano
  - Nara, Nara
  - Ōita, Oita Prefecture
  - Kurashiki-shi, Okayama-ken
  - Okayama, Okayama-ken
  - Hirakata-shi, Osaka
  - Ibaraki-shi, Osaka
  - Ikeda-shi, Osaka
  - Osaka, Osaka
  - Sakai-shi, Osaka
  - Suita-shi, Osaka
  - Tondabayashi-shi, Osaka
  - Toyonaka-shi, Osaka
  - Iruma-shi, Saitama
  - Kusatsu-shi, Shiga
  - Hamamatsu, Shizuoka
  - Numazu-shi, Shizuoka
  - Yaizu-shi, Shizuoka
  - Komatsushima-shi, Tokushima
  - Naruto-shi, Tokushima
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Machida-shi, Tokyo
  - Minato-ku, Tokyo
  - Ohta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Suginami-ku, Tokyo
  - Toyama, Toyama
  - Yamaguchi, Yamaguchi

REFERENCES:
- [Derived] Osuga Y, Seki Y, Tanimoto M, Kusumoto T, Kudou K, Terakawa N. Relugolix, an oral gonadotropin-releasing hormone receptor antagonist, reduces endometriosis-associated pain in a dose-response manner: a randomized, double-blind, placebo-controlled study. Fertil Steril. 2021 Feb;115(2):397-405. doi: 10.1016/j.fertnstert.2020.07.055. Epub 2020 Sep 7. PMID 32912633